CLINICAL TRIAL: NCT05379153
Title: The Revitalize Trial: Reducing Vaginal Atrophy With Fractional CO2 Laser for Breast Cancer Survivors
Brief Title: Testing Laser Therapy for Treatment of Vaginal Dryness in Survivors of Breast Cancer, The Revitalize Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221801; NCI-2022-02754 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Vaginal Atrophy
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The provider will not be blinded to the arm the patient is on. PRO measures will be administered by research personnel who are blinded to the arm the patient is enrolled on at each study time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (vaginal fractional CO2 laser therapy) (Experimental): Patients undergo vaginal fractional CO2 laser therapy over 20-30 minutes every 6 weeks for 3 treatments in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Laser Therapy; Other: Questionnaire Administration; Other: Quality of Life Assessment
- Arm II (placebo) (Sham Comparator): Patients undergo placebo procedure over 20-30 minutes every 6 weeks for 3 treatments in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Sham Intervention; Other: Questionnaire Administration; Other: Quality of Life Assessment

INTERVENTIONS:
Device: Laser Therapy — Undergo vaginal fractional CO2 laser therapy
  Arms: Arm I (vaginal fractional CO2 laser therapy)
Device: Sham Intervention — Undergo placebo procedure
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies
Other: Quality of Life Assessment — Ancillary studies

SUMMARY:
This phase III trial tests whether vaginal fractional CO2 laser therapy works in treating vaginal dryness in breast cancer survivors. Vaginal dryness can be commonly experienced with normal aging, with menopause, or come about from medications used to treat breast cancer such as chemotherapy or endocrine therapies like tamoxifen or aromatase inhibitors. Vaginal fractional CO2 laser therapy may help reduce vaginal dryness.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether vaginal fractional carbon dioxide (CO2) laser treatment is superior to vaginal placebo procedure in improving the severity of vaginal dryness, based on an 11-point (0-10) patient reported numerical analog scale.

SECONDARY OBJECTIVES:

I. To determine whether vaginal fractional CO2 laser treatment is superior to vaginal placebo procedure in improving patient-reported vaginal discomfort during sexual activity, based on the vaginal discomfort domain of the Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function version (v.) 2.0 Brief Profile-Female.

II. To determine whether vaginal fractional CO2 laser therapy results in improvement in patient-reported quality of life, based on a single item 11-point numerical analog scale.

III. To evaluate potential toxicities associated with vaginal fractional CO2 laser therapy.

OUTLINE: Patients are randomized at a 2:1 ratio to Arm I and Arm II.

ARM I: Patients undergo vaginal fractional CO2 laser therapy over 20-30 minutes every 6 weeks for 3 treatments in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo placebo procedure over 20-30 minutes every 6 weeks for 3 treatments in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks, and 3,6, 12, 18 and 24 months after the last procedure visit.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of breast cancer treated with curative intent who have completed primary therapy (consisting of surgery with or without chemotherapy, targeted therapy, immunotherapy and/or radiation) >= 12 months prior to registration. Concurrent trastuzumab /pertuzumab is permissible
* May be receiving ongoing adjuvant endocrine therapy (with an AI or tamoxifen +/- ovarian function suppression). Patients are not required to receive these treatments to be eligible. Participants receiving adjuvant endocrine therapy prior to registration must intend to continue the same endocrine therapy for the 4 months while they are receiving protocol treatment, unless a clinically necessary change is indicated at the discretion of the patient's medical oncologist. Patients on aromatase inhibitor (AI) therapy, tamoxifen with or without ovarian function suppression therapy must have been on their current endocrine therapy regimen for at least 6 months prior to registration
* Patient-reported vaginal dryness with or without dyspareunia of at least moderate severity on average, defined as >= 4 on a 0-10-point scale that has been bothersome for >= 3 months and for which the patient wants to undergo the study procedure
* No evidence of metastatic breast cancer. Scans to assess for metastatic disease are not required for eligibility
* No prior gynecologic cancer, vaginal intra-epithelial neoplasia, pelvic radiation or pelvic reconstructive surgery utilizing mesh. Patients with cervical intraepithelial neoplasia are eligible
* No history of scleroderma, lupus, systemic sclerosis, mixed connective tissue disorder, undifferentiated connective tissue disorder or collagen vascular disease, dermatomyositis, polymyositis, lichen sclerosis or vulvar vestibulitis
* No pelvic surgery that involved a vaginal incision within 6 months of registration. Patients who received laparoscopic BSO (Bilateral salpingooophorectomy) are eligible
* No systemic estrogen or progesterone, vaginal estrogen, vaginal prasterone, ospemifene, and/or androgen therapy within 6 weeks prior to registration
* No other suspected contraindications for undergoing laser therapy
* No prior vaginal laser therapy at any time. Patients who would have completed any type of vaginal laser resurfacing procedure at any time prior to the start of study treatment are not eligible
* No known concurrent invasive carcinoma/malignancy. Patients with carcinoma in situ are eligible. Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible if not currently receiving treatment
* Postmenopausal based on at least one of the following criteria at the time of registration:

  * Women 50 or older with no spontaneous regular menses > 12 months
  * On ovarian suppression (i.e., gonadotrophin releasing hormone [GNRH] agonist/antagonist) for at least 6 months or greater, with plans to continue such treatment for at least 18 weeks
  * Bilateral oophorectomy
  * Women on AI therapy (i.e., clinically judged to be postmenopausal)
* In order to complete the mandatory patient-completed measures, participants must be able to speak, read and understand English or Spanish
* Age >= 22 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* No medical history of: keloid formation, genital fistula, thin recto-vaginal septum (defined as a distance of < 2 cm between the vaginal opening and the anal opening)

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Changes in patient reported vaginal dryness severity | Up to 18 weeks
  Will use an 11-point (0-10) numerical analog scale to assess patient reported severity of vaginal dryness. Higher scores represent worse symptoms (0: None - 10: Worst possible). The vaginal dryness scores at each time point will be summarized separately by treatment arm using the mean (standard deviation) and median (range). The score changes from baseline to the 18-week time point (T4) will be compared using two-sample t-test or Wilcoxon rank-sum test as appropriate.

SECONDARY OUTCOMES:
Changes in vaginal discomfort during sexual activity (for sexually active subset of study population only) | Baseline up to 24 months after completion of treatment
  Assessed using the Vaginal discomfort domain of Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function version (V) 2.0 Brief Profile - Female (only the sexually active women will be evaluable for this, which is estimated to be approximately 50% of the population). Higher scores represent more discomfort (1: None - 5: A lot). Change in the vaginal discomfort domain of the PROMIS Sexual Function v. 2.0 Brief Profile-Female from baseline to each post-therapy-initiation time point will be summarized by treatment arm and will be compared as described for the primary endpoint.
Change in quality of life | Baseline up to 24 months after completion of treatment
  Evaluated using 11-point (0-10) numerical analog scale. Higher scores represent better quality of life (0: As bad as it can be - 10: As good as it can be). Change in patient reported quality of life from baseline to each post-therapy initiation time point will be summarized and compared as described for the primary endpoint.
Incidence of adverse events associated with vaginal fractional CO2 laser therapy | Up to 24 months after completion of treatment
  Incidences of toxicities in the fractional CO2 laser therapy arm will be summarized by type. Common toxicities that occur in both arms will be summarized and compared between arms using the Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Lustberg, MD, MPH, Study Chair — Yale University Comprehensive Cancer Center